CLINICAL TRIAL: NCT05346497
Title: Surgical Management of the Aortic Root and Long-term Outcomes For Acute Type A Aortic Dissection
Status: Completed | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2021-776R
Record Dates: First submitted 2022-01-21; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Type A Aortic Dissection
Keywords: Type A Aortic Dissection; Aortic Root Surgery
MeSH Terms: interventions — Red Cross

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Bentall: Patients who underwent Bentall procedure for ATAAD
  Interventions: Procedure: Bentall
- David: Patients who underwent David procedure for ATAAD
  Interventions: Procedure: David
- ARR: Patients who underwent aortic root reconstruction procedure except Bentall and David procedure for ATAAD
  Interventions: Procedure: ARR

INTERVENTIONS:
Procedure: Bentall — Bentall procedure: include replacement of both aortic valve and root
  Groups: Bentall
Procedure: David — David procedure: include replacement of aortic root and aortic valvuloplasty
  Groups: David
Procedure: ARR — Aortic root reconstruction: reconstruction instead of replacement of aortic root, without surgery of the valve. include sandwich procedure, adventitia invertion procedure, etc.
  Groups: ARR

SUMMARY:
The investigators focus on the patients who underwent aortic root surgery for acute type A aortic dissection between 2005.01-2021.11. The patients are divided into 3 groups according to the different aortic root surgical methods(Bentall，David and root reconstruction). Clinical data including age, gender, comorbidities, surgical informations and perioperative informations will be collected. All patients will receive follow-ups in hospital or by telephone.

All the informations will be analyzed by SPSS to show the difference of both perioperative and long-term results among different surgical strategies.

DETAILED DESCRIPTION:
Acute type A aortic dissection (ATAAD) is a rare but life threatening situation requiring immediate intervention. Regarding emergency operation for ATAAD, an important principle is to reconstruct the afflicted aorta to prevent fatal rupture.

For aortic root dissection, the Bentall procedure has been the standard operation and has been proven simple and effective. However, the requirement for lifelong anticoagulation therapy is associated with increased risk of thromboembolic and bleeding complications. Valve sparing aortic root reimplantation (David reimplantation), which has been proven effective in root aneurysm with satisfactory safety and long-term outcomes, is an appealing alternative to preserve native aortic valve, especially for younger patients with intact valve function. Aortic root reconstruction without valve surgery is also a well-used strategy for aortic root dissection, but the long-term outcome is still controversial.

The investigators focus on the patients who underwent aortic root surgery for acute type A aortic dissection between 2005.01-2021.11. The patients are divided into 3 groups according to the different aortic root surgical methods(Bentall，David and root reconstruction). Clinical data including age, gender, comorbidities, surgical informations and perioperative informations will be collected. All patients will receive follow-ups in hospital or by telephone.

All the informations will be analyzed by SPSS to show the difference of both perioperative and long-term results among different surgical strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were followed up at our hospital for aortic lesions or who underwent aortic root surgery (including the Bentall procedure, the David procedure, and other aortic root angioplasty or replacement procedures)
* Patients older than 18 years of age, no specific gender requirement
* Patients who are compliant and able to complete follow-up
* Patients who understand the purpose of the study, voluntarily participate, and have signed the Biospecimen and Health-Related Information Donation Form by themselves or their legal representative.
* Patients who understand the purpose of the study, voluntarily participate and have signed the informed consent form for donation of biological samples and health-related information by themselves or their legal representative

Exclusion Criteria:

* Patients who are unable or unwilling to participate in the study and sign the informed consent form
* Patients with poor compliance and unable to complete follow-up
* Patients with severe organ insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Based on currently available data on aortic-related procedures in our department from 2005 to 2021, we expect to include 1600 patients at the end of the study.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Death for any reason | From date of surgery until the date of death for any reason, up to 20 years
  Death for any reason

SECONDARY OUTCOMES:
Redo aortic surgery | From date of surgery until the date of redo aortic surgery for any reason, up to 20 years
  Patients underwent aortic surgery again for any reason

IPD SHARING:
Plan to Share IPD: Undecided